CLINICAL TRIAL: NCT06526663
Title: Randomizing Vignettes to Understand Contributors to Trust in Primary Care Doctors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00447825; K24AG049036 (NIH)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Primary Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Vignette1 (Active Comparator): abbb
  Interventions: Behavioral: vignette exposure
- Vignette2 (Active Comparator): aabb
  Interventions: Behavioral: vignette exposure
- Vignette3 (Active Comparator): aaab
  Interventions: Behavioral: vignette exposure
- Vignette4 (Active Comparator): aaaa
  Interventions: Behavioral: vignette exposure
- Vignette5 (Active Comparator): babb
  Interventions: Behavioral: vignette exposure
- Vignette6 (Active Comparator): baab
  Interventions: Behavioral: vignette exposure
- Vignette7 (Active Comparator): baaa
  Interventions: Behavioral: vignette exposure
- Vignette8 (Active Comparator): abaa
  Interventions: Behavioral: vignette exposure
- Vignette9 (Active Comparator): abba
  Interventions: Behavioral: vignette exposure
- Vignette10 (Active Comparator): bbab
  Interventions: Behavioral: vignette exposure
- Vignette11 (Active Comparator): bbaa
  Interventions: Behavioral: vignette exposure
- Vignette12 (Active Comparator): bbba
  Interventions: Behavioral: vignette exposure
- Vignette13 (Active Comparator): bbbb
  Interventions: Behavioral: vignette exposure
- Vignette14 (Active Comparator): baba
  Interventions: Behavioral: vignette exposure
- Vignette15 (Active Comparator): abab
  Interventions: Behavioral: vignette exposure
- Vignette16 (Active Comparator): aaba
  Interventions: Behavioral: vignette exposure

INTERVENTIONS:
Behavioral: vignette exposure — Participants will be randomized to be exposed to one of 16 written vignettes that vary four elements of the primary care experience. The four attributes can take two levels.
  In the second round, individuals will be randomized to only 4 different vignettes.

SUMMARY:
In this proposed work, the investigators plan to generate experimental evidence about trust and overuse of healthcare. The protocol described below is for the first phase of this work to establish the feasibility of modifying feelings of trust via a vignette.

DETAILED DESCRIPTION:
The investigators will engage survey participants by recruiting from among the "Workers" registered with Amazon Mechanical Turk (MTurk). These are paid participants who chose to participate in this anonymous, low-risk activity. After pilot testing on a small set of Workers, the investigators will field the full survey using a randomized design to test hypotheses about the investigators ability to manipulate trust experimentally.

Individuals eligible as participants will be over the age of 18 years, able to read and respond in English, and have had one or more visits with a doctor in the past 3 years.

Survey

The survey has three parts. The investigators will use Qualtrics to develop the survey vignette and use the randomization feature of Qualtrics to randomize the participants when the participant clicks on the link to Qualtrics.

1. Vignette Participants will be randomized to view one of sixteen vignettes. The vignettes describe a clinical encounter and vary four attributes, each of which has two levels.

   Duration of relationship with doctor: No previous relationship (episodic care, walk-in-care, on demand telemedicine) versus > 3 years; Connection: Physician is attending to computer versus Physician is attending to patient; Length of visit: 15 minutes versus 30 minutes; Shares information: Doctor does not explain the decision making versus Doctor shares what he/she knows that informed the decision

   A sample vignette is presented here:

   Imagine having low back pain that started 4 days ago and being very uncomfortable. For this visit, the patient sees a doctor at the usual practice that the patient has never met before. The doctor spends 30 minutes with the patient. He is primarily looking at the computer screen and not at the patient. At the end, the doctor tells the patient that no xrays are needed and makes recommendations for treating the patient's pain.

   The investigators will do a test of attention quiz to assure that the participant read the vignette asking:
   1. Why did you go for care? (twisted ankle, back pain)
   2. Did the doctor make any recommendations? (recommended pain treatment, recommended a cast)
2. Trust in Clinician Survey.

The investigators will use the Wake Forest Trust in Physician (WFTP) scale slightly modified to clarify that the investigators are inquiring about the clinician described in the vignette. Whereas the WFTP scale asks about "your doctor", the investigators will ask about "this doctor". The WFTP uses a 5-pt Likert scale. Items 2, 3, and 8 are reverse coded upon analysis (strongly agree, agree, neutral, disagree, strongly disagree).

The introduction will read:

Think about the visit described above. What do you think about this doctor?

1. This doctor will do whatever it takes to get you all the care you need.
2. Sometimes this doctor cares more about what is convenient for [him or her] than about the patient's medical needs.
3. This doctor's medical skills are not as good as they should be.
4. This doctor is extremely thorough and careful.
5. You completely trust this doctors decisions about which medical treatments are best for you.
6. This doctor is totally honest in telling you about all of the different treatment options available for the patient's condition.
7. This doctor only thinks about what is best for you.
8. Sometimes this doctor does not pay full attention to what you are trying to tell [him or her].
9. The patient has no worries about putting the patient's life in this doctor's hands.
10. All in all, the patient has complete trust in this doctor.

3) Demographics

The investigators will ask the respondents to describe themselves as follows:

Sex (Male, Female, Non-binary) Age (18-35, 36-50, 51-65, >=65) Race/Ethnicity (Black, White, Asian, Native American/Pacific Islander, Hispanic, Other) Choose all that apply How do you describe your health? Excellent, Very good, Good, Fair, Poor Do you have health insurance? Yes or No What is your highest level of education completed? Grade school, High School, college, post-graduate

Analysis The investigators will use descriptive statistics to describe the characteristics of the respondents and the distribution of the WFTP score, which is a quasi-continuous measure. The investigators will look for outliers defined as scores greater or less than 3.2 standard deviations from the mean. Linearity will be examined with scatterplots. The assumption of normality will be assessed by analyzing the skewness and kurtosis of the variables and with use of histograms. The investigators expect the WFTP to be normally distributed as it has been in other populations. If it is not, the investigators will consider log transformation. The investigators will describe the respondents by vignette assignment to confirm that randomization was successful.

Given the structure of MTurk, the investigators will not have a measure of survey response. The investigators will, however, be able to assess the pattern of missing variables across the responses and will incorporate this appropriately into the models.

In the validation study by Katz, she reports in a national sample, the Wake Forest Physician Trust Scale (WFPTS) had a mean score of 40.8 (SD = 6.2) for the national sample of 959 participants. In her study of fewer participants recruited from MTurk, the mean score for the WFPTS was 35.9 (SD = 6.12) for young adult participants and 36.1 (SD = 6.11) for older adult participants.

The investigators would like to be able to detect a 2 standard deviation (SD) difference between the lower trust vignettes and the higher trust vignettes. If the study has 36 individuals in each group, the investigators are able to detect, with a power of 0.8 and an alpha of 0.5, a difference of 4 points on the WFTP (38 (sd 6) vs 42 (sd 6)). The investigators will aim to have 36 respondents in each of 16 groups.

The investigators will test hypotheses about the vignettes and the reported trust in the physician.

For the second round of the survey, investigators will randomize to only 4 arms depending on the results of the first round. The investigators will randomize 100 individuals (50 men and 50 women) to each of the 4 arms.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be over the age of 18 years,
* able to read and respond in English, and
* have had one or more visits with a doctor in the past 3 years
* will be registered MTURK workers

Exclusion Criteria:

* None

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self identified women and men or non-binary individuals are eligible
Enrollment: 1106 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Wake Forest Physician Trust Scale (10 item survey) | Immediately upon completing exposure to the vignette
  Scores range from 10-50 with higher scores indicating higher trust

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Segal, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Virginia Tech, Blacksburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data without identifiers will be shared upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years after collection
Access Criteria: Data will be shared for non-commercial purposes that are reasonable requests.